CLINICAL TRIAL: NCT05091255
Title: Cryotherapy in the Treatment of Desmoid Tumors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Principal Investigator, Costantino Errani, Principal Investigator, Istituto Ortopedico Rizzoli
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRYODESMO
Record Dates: First submitted 2021-10-12; First posted 2021-10-25 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Desmoid
Keywords: desmoid tumor; cryotherapy
MeSH Terms: conditions — Desmoid Tumors | interventions — Cryotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients (Experimental)
  Interventions: Procedure: Cryotherapy

INTERVENTIONS:
Procedure: Cryotherapy — The procedure involves general or peripheral anesthesia and percutaneous treatment under CT control with probes capable of forming ice spheres of up to 3 cm that will be used in sufficient number to treat the neoplasm completely.

SUMMARY:
Desmoid tumor is a benign neoplasm with an unpredictable course and a high rate of local recurrence if treated surgically. Therefore, over time the surgical approach has become conservative, preferring simple observation or medical therapy in case of disease progression through the use of hormonal therapy and low-dose chemotherapy. Since this neoplasm remains benign, our study aims to avoid chemotherapy in patients usually young through the use of a minimally invasive treatment such as cryotherapy.

ELIGIBILITY:
Inclusion Criteria:

* histologic diagnosis of desmoid tumors
* age > 18 years
* abdominal and extra-abdominal desmoid tumors

Exclusion Criteria:

* contraindication to the procedure by the interventional radiologist in terms of tumor proximity to neurologic/vascular structures
* retroperitoneal desmoid tumors
* age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2021-05-20 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
response to treatment | At baseline (time 0)
  assessment of tumor response to treatment will be performed using the solid tumor response criteria

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Itituto Ortopedico Rizzoli, Bologna, BO, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kujak JL, Liu PT, Johnson GB, Callstrom MR. Early experience with percutaneous cryoablation of extra-abdominal desmoid tumors. Skeletal Radiol. 2010 Feb;39(2):175-82. doi: 10.1007/s00256-009-0801-z. Epub 2009 Sep 21. PMID 19768644
- [Background] Redifer Tremblay K, Lea WB, Neilson JC, King DM, Tutton SM. Percutaneous cryoablation for the treatment of extra-abdominal desmoid tumors. J Surg Oncol. 2019 Sep;120(3):366-375. doi: 10.1002/jso.25597. Epub 2019 Jun 24. PMID 31236956
- [Background] Schmitz JJ, Schmit GD, Atwell TD, Callstrom MR, Kurup AN, Weisbrod AJ, Morris JM. Percutaneous Cryoablation of Extraabdominal Desmoid Tumors: A 10-Year Experience. AJR Am J Roentgenol. 2016 Jul;207(1):190-5. doi: 10.2214/AJR.15.14391. Epub 2016 Apr 11. PMID 27064168